CLINICAL TRIAL: NCT05083650
Title: Comparison of Macular Hole Closure Rate in Patients With Poor Prognosis Clinical Features Treated With Amniotic Membrane Graft With and Without Limitorrhexis
Brief Title: Large Macular Hole Closure Rate With Amniotic Membrane Graft With and Without Limitorrhexis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Principal Investigator, Jose Luis Rodriguez Loaiza, Medical Subdirector, Instituto de Oftalmología Fundación Conde de Valenciana
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: MAM CONDE
Record Dates: First submitted 2019-06-25; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Macular Holes
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Intervention Model Description: Large MHs (diameter > 550 μm)
Who Masked: Participant, Care Provider
Masking Description: We never let the patient know the performed surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amniotic membrane without internal limiting membrane peeling (Experimental): The surgery performed will be phacoemulsification + vitrectomy using an amniotic membrane to plug the macular hole using air as tamponade.
  Interventions: Procedure: Macular hole closure with amniotic membrane with/without internal limiting membrane peeling
- Amniotic membrane with internal limiting membrane peeling (Active Comparator): The surgery performed will be phacoemulsification + vitrectomy + internal limiting membrane peeling using an amniotic membrane to plug the macular hole using air as tamponade.
  Interventions: Procedure: Macular hole closure with amniotic membrane with/without internal limiting membrane peeling

INTERVENTIONS:
Procedure: Macular hole closure with amniotic membrane with/without internal limiting membrane peeling — Pars plana vitrectomy with/without internal limiting membrane peeling, amniotic membrane, and air tamponade

SUMMARY:
Patients with idiopathic macular holes (MHs) postoperative closure rates for large MHs (diameter > 550 μm) are disappointing and often require a second intervention, different techniques have been described with very variable success rates in different published studies, an efficient technique with good functional outcome has not been found.

DETAILED DESCRIPTION:
Interventional study in large macular holes (diameter > 550 μm) using an amniotic membrane with and without internal limiting membrane peeling.

ELIGIBILITY:
Inclusion Criteria:

* Not myopic patients (<6 Dioptre or <26 mm)
* Large macular hole >550 μm
* > 6 months symptoms
* Signing informed consent

Exclusion Criteria:

* Patients with other ocular disease (diabetic retinopathy, glaucoma, uveitis, ocular tumors, etc)
* Using systemic drugs that are toxic for the optic nerve or retina (chloroquine, hydroxychloroquine, tamoxifen, ethambutol, etc)
* Patients with ocular surgery

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-03-10 (Estimated)

PRIMARY OUTCOMES:
% of macular hole clousure measured with OCT | 6 months
  Closure of the macular hole by optical coherence tomography

SECONDARY OUTCOMES:
Best-corrected visual acuity measured with Snellen Chart | 6 months
  Improvement of 2 lines in best-corrected visual acuity
Superficial and deep retinal capillary plexus density with OCT-A | 6 months
  Presence of capillary plexus in macular hole area

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rios Esquer, MD, Principal Investigator — Instituto de Oftalmologia Conde de Valenciana; Ishtar A Astorga Carballo, MD, Principal Investigator — Instituto de Oftalmologia Conde de Valenciana; Jose L Rodriguez Loaiza, MD, Principal Investigator — Instituto de Oftalmologia Conde de Valenciana; Zita Chao Loyo, MD, Principal Investigator — Instituto de Oftalmologia Conde de Valenciana; Felipe Esparza Correa, MD, Principal Investigator — Instituto de Oftalmologia Conde de Valenciana
Locations (1):
- Instituto de Oftalmologia Conde de Valenciana, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided